CLINICAL TRIAL: NCT04582981
Title: A Randomized, Controlled Phase II Clinical Trial of Fruquintinib Combined With Raltitrexed Versus Fruquintinib Monotherapy in Patients With Advanced Colorectal Cancer Who Had Failed Second-line or Above Standard Chemotherapy
Brief Title: Fruquintinib and Raltitrexed Versus Fruquintinib Monotherapy in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Weijian Guo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-FRaF
Record Dates: First submitted 2020-10-03; First posted 2020-10-12 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Advanced Colorectal Carcinoma
Keywords: advanced colorectal cancer; fruquintinib; raltitrexed; target therapy
MeSH Terms: interventions — HMPL-013; raltitrexed

STUDY DESIGN:
Intervention Model Description: This study is an open-label, randomized, controlled, multi-centered phase II clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Combination treatment of Fruquintinib and Raltitrexed
  Interventions: Drug: Fruquintinib and raltitrexed
- Arm B (Experimental): Monotherapy of Fruquintinib
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib and raltitrexed — Fruquintinib 5mg qd plus raltitrexed 2mg/m2, q2w
  Other Names: F and R
  Arms: Arm A
Drug: Fruquintinib — Fruquintinib 5mg qd monotherapy
  Other Names: F
  Arms: Arm B

SUMMARY:
A randomized, controlled phase II clinical trial of Fruquintinib combined with Raltitrexed versus Fruquintinib monotherapy in patients with advanced colorectal cancer who had failed second-line or above standard chemotherapy

DETAILED DESCRIPTION:
This study plans to evaluate the clinical benefits of fruquintinib combined with raltitrexed compared with fruquintinib single drug treatment in patients with advanced colorectal cancer who have failed second-line or above treatment, in order to explore the rationality of this strategy with chemotherapy + targeted combination therapy and obtain the relevant survival and safety data. A total of 136 patients were planned to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. no less than 18 years old
2. confirmed by histopathological examination, recurrent/metastatic colorectal adenocarcinoma
3. had received at least two lines standard chemotherapy and failed. These standard regimens must include fluorouracil, oxaliplatin, and irinotecan. Treatment failure was defined as disease progression within 3 months after the last treatment or intolerance of toxicity or side effects during treatment ; Note: A. each line of treatment shall include more than one cycle of chemotherapeutic agents; B. adjuvant/neoadjuvant therapy is allowed in the former treatment. If recurrence or metastasis occurs during adjuvant/neoadjuvant therapy or within 6 months after completion, adjuvant/neoadjuvant therapy is considered a failure of first-line chemotherapy for the advanced disease; C. Prior antitumor therapy regimens using chemotherapy combined with cetuximab or bevacizumab were permitted.
4. with one or more measurable lesions, according to RECIST criteria, version 1.1;
5. Eastern Cooperative Oncology Group (ECOG) performance score(PS) from 0 to 2;
6. Life expectancy no less than 12 weeks;
7. Acceptable hematologic, hepatic, and renal function within 7 days from screening： the blood neutrophil count≥1.5x109 /L; hemoglobin ≥ 9.0 g/dl，the blood platelet count≥80 x109 /L, total bilirubin < 1.5 x upper normal limit（UNL), alanine aminotransferase（ALT） and aspartate transaminase（AST）< 2.5 x UNL(< 5 x UNL for patients with live metastasis), serum creatinine≤1 x UNL，endogenous creatinine clearance rate >50ml/min
8. Women of reproductive age need to take effective contraceptive measures.
9. Participate in this study voluntarily and sign informed consent. Understand the purpose of this study and the necessary procedures. Good compliance to cooperate with the follow-up.

Exclusion Criteria:

1. urine protein 2 + or above, or 24 hours urinary protein quantitative acuity 1.0 g / 24 h
2. Abnormal coagulation function or those receiving thrombolytics or anticoagulants
3. Patients with tendency of gastrointestinal hemorrhage, including active peptic ulcer with fecal occult blood ++, hematemesis or melena within 3 months
4. Received other systemic anti-tumor therapy, including cell signal transduction inhibitors, drug therapy, immune therapy within 3 weeks
5. With uncontrolled high blood pressure (systolic blood pressure > 140 MMHG, diastolic blood pressure > 90 MMHG)
6. Radiotherapy therapy for target lesions
7. symptomatic cerebral or meningeal metastasis;
8. Uncontrolled pleural or peritoneal effusion
9. Undergoing dialysis
10. Severe or uncontrolled infection
11. With multiple factors that affecting oral administration
12. Former exposed to any VEGFR tyrosine kinase inhibitors (e.g regorafenib, apatinib, anlotinib etc.) for treatment
13. Raltitrexed treatment for more than one cycle in former line therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | assessed up to 24 months
  the time from randomization to tumor progression or death from any cause,whichever came first

SECONDARY OUTCOMES:
overall survival (OS) | assessed up to 36 months
  the time from randomization to death from any cause,whichever came first,
objective response rate (ORR) | through study completion, an average of 2 year
  The proportion of patients whose tumors shrink to a certain extent and remain constant for a certain period of time
disease control rate (DCR) | through study completion, an average of 2 year
  Percentage of cases with response to treatment (PR+CR) and disease stability (SD) that can be evaluated

OTHER OUTCOMES:
quality of life score (QOL) | through study completion, an average of 2 year
  EORTC QOL-C30, version 3.0,

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Result] Pfeiffer P, Yilmaz M, Moller S, Zitnjak D, Krogh M, Petersen LN, Poulsen LO, Winther SB, Thomsen KG, Qvortrup C. TAS-102 with or without bevacizumab in patients with chemorefractory metastatic colorectal cancer: an investigator-initiated, open-label, randomised, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):412-420. doi: 10.1016/S1470-2045(19)30827-7. Epub 2020 Jan 27. PMID 31999946
- [Result] Cunningham D, Zalcberg JR, Rath U, Oliver I, van Cutsem E, Svensson C, Seitz JF, Harper P, Kerr D, Perez-Manga G. Final results of a randomised trial comparing 'Tomudex' (raltitrexed) with 5-fluorouracil plus leucovorin in advanced colorectal cancer. "Tomudex" Colorectal Cancer Study Group. Ann Oncol. 1996 Nov;7(9):961-5. doi: 10.1093/oxfordjournals.annonc.a010800. No abstract available. PMID 9006748